CLINICAL TRIAL: NCT04512274
Title: A Single Center Study in 22 Healthy Male and Female Subjects to Investigate the Skin Protectant and Anti-Inflammatory Properties of Omeza Collagen Matrix on Damaged Skin
Brief Title: Skin Protectant Properties of Omeza Collagen Matrix on Damaged Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OMZIFL3M
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Transepidermal Water Loss; Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Test Article (Experimental): The test article was applied to an open application site and to a second site of induced inflammation
  Interventions: Device: Test Article

INTERVENTIONS:
Device: Test Article — Omeza Collagen Matrix

SUMMARY:
Single-blind within subject comparison study conducted to investigate the skin protectant properties of Omeza Collagen Matrix on damaged skin

DETAILED DESCRIPTION:
This study was conducted in 22 healthy subjects to determine the skin protectant and anti-inflammatory properties of the test product.

For the skin protectant assay the test article was applied to the forearm and covered with gauze for 10 minutes before assessment of irritation and TEWL readings.

An inflammatory skin response was induced by a SLS solution 24 hours prior to application of the test article. The test article was applied for 10 minutes at the site of inflammation. The test site was then graded for irritation and TEWL readings.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female, aged 18 years or older.
* Subject has signed a written Informed Consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Inadequate precaution or procedure to prevent pregnancy (women of child bearing potential only).
* A current skin disease of any type at the test site (e.g. eczema, psoriasis)
* Heavy alcohol consumption in the opinion of the investigator.
* A fever in the last 12 hours, prior to the initial patch application.
* Significant past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, locomotor or psychiatric disease, which in the opinion of the Investigator would compromise the safety of the subject.
* History of malignant disease.
* Insulin dependent or non-insulin dependent diabetes.
* Concurrent medication likely to affect the response to the test articles or confuse the results of the study, i.e. routine high dosage use of antiinflammatory drugs (aspirin, ibuprofen, corticosteroids).
* Known sensitivity to the treatment solutions or their constituents including patch materials.
* Sensitisation or questionable sensitisation in a Repeat Insult Patch Test.
* Use of self-tanning lotion on the test area, one week previous to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Transepidermal Water Loss (TEWL) | 24 hours
  Assessment of water evaporation (TWEL) based upon diffusion principle after 24 hour injury
Transepidermal Water Loss (TEWL) | 48 hours
  Assessment of water evaporation (TWEL) based upon diffusion principle
Transepidermal Water Loss (TEWL) | 72 hours
  Assessment of water evaporation (TWEL) based upon diffusion principle
Transepidermal Water Loss (TEWL) | 96 hours
  Assessment of water evaporation (TWEL) based upon diffusion principle

SECONDARY OUTCOMES:
Erythema | 24 hours
  Irritancy Grading on a 0-4 scale
Erythema | 48 hours
  Irritancy Grading on a 0-4 scale
Erythema | 72 hours
  Irritancy Grading on a 0-4 scale
Erythema | 96 hours
  Irritancy Grading on a 0-4 scale

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Drewitt, Principal Investigator — PCR Corp; Andrew King, Study Director — PCR Corp
Locations (1):
- Princeton Research Corporation, Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No